CLINICAL TRIAL: NCT03097900
Title: Does Caffeine Enhance Bowel Recovery After Colorectal Surgery?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFFEINE-HMO-CTIL
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Ileus
Keywords: Postoperative Ileus; Caffeine Citrate
MeSH Terms: interventions — caffeine citrate; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Caffeine Citrate) group (Active Comparator): 25 patients after elective colorectal surgery will be given 100 mg caffeine citrate orally diluted in 50 ml apple flavored water three times per day starting on the morning of postoperative day 1 after surgery until flatus will occur for the first time or to a maximal period time of 7 days, whichever comes earlier.
  Interventions: Drug: Caffeine Citrate
- Placebo (Water) group (Placebo Comparator): 25 patients after elective colorectal surgery will be given 50 ml apple flavored water three times per day starting on the morning of postoperative day 1 after surgery until flatus will occur for the first time or to a maximal period time of 7 days, whichever comes earlier.
  Interventions: Other: Water

INTERVENTIONS:
Drug: Caffeine Citrate — 25 patients after elective colorectal surgery will be given 100 mg caffeine citrate orally diluted in 50 ml apple flavored water three times per day starting on the morning of postoperative day 1 after surgery until flatus will occur for the first time or to a maximal period time of 7 days, whichever comes earlier.
  Other Names: Cafcit
  Arms: Treatment (Caffeine Citrate) group
Other: Water — 25 patients after elective colorectal surgery will be given 50 ml apple flavored water three times per day starting on the morning of postoperative day 1 after surgery until flatus will occur for the first time or to a maximal period time of 7 days, whichever comes earlier.
  Arms: Placebo (Water) group

SUMMARY:
Postoperative ileus is a frequently occurring surgical complication. It is defined as temporary inhibition of propulsive bowel activity and is manifested by abdominal distention, nausea, vomiting and diet intolerance. It may lead to a prolonged hospital stay, hospital-acquired infections or complications that may require additional treatments (e.g. analgesia, fluids, electrolyte replacement, nasogastric tube decompression), and as a result increase medical costs.

Previous studies showed that postoperative coffee consumption shortens the time to first bowel movement after colorectal resections. However, none could explain the mechanism by which coffee stimulates intestinal motility and the determinant agent for this action is still up for discussion (either caffeine or another coffee component).

Coffee has a negligible caloric content; It has a pH that varies from 5 to 6 (less acidity than other beverages that have no similar effect on bowel motility) and it is hypotonic. Therefore, it is highly unlikely that bowel motility is due to the physical properties of the coffee. Much more likely, that one (or more) of the numerous phytochemicals of the coffee bean are responsible for this effect, when the most obvious candidate seems to be caffeine. However, as mentioned above, very little evidence exists that caffeine was responsible for the observed effect on colonic function in previous studies.

The purpose of this single-centered, prospective, single blinded, randomized clinical trial is to evaluate whether the use of caffeine in the post-operative period significantly reduces the duration of postoperative ileus, and therefore, improves recovery and shorten the hospital stay.

The study hypothesis is that post-operative use of caffeine will reduce time to recovery of GI function (post-operative ileus) by at least 15 hours and thus reduce hospital length of stay by at least 15 hours in patients undergoing elective colorectal operations.

50 patients due to undergo large bowel resection via laparotomy or laparoscopy will be enrolled and randomized (1:1) to those who will receive caffeine (100 mg 3 times per day) and those who will receive placebo (tap water) starting on the morning of postoperative day 1 after surgery until flatus will occur for the first time or to a maximal period time of 7 days, whichever comes earlier.

DETAILED DESCRIPTION:
Background Postoperative ileus is a frequently occurring surgical complication. It is defined as temporary inhibition of propulsive bowel activity and is manifested by abdominal distention, nausea and vomiting and diet intolerance. It may lead to a prolonged hospital stay, hospital-acquired infections or complications that may require additional treatments (analgesia, intravenous fluid administration, electrolyte replacement, nasogastric tube decompression etc.) and as a result increase medical costs.

Surgeons are continually trying to find ways to shorten postoperative ileus. The means are diverse and include advancing diet as tolerated, avoiding the use of nasogastric tubes, early ambulation, occasional use of gastrograffin or alvimopan (a selective μ-receptor opioid antagonist) and the use of minimally invasive surgery (laparoscopic colectomy) rather than laparotomy. Asao et al showed that chewing gum after laparoscopic colectomy leads to an earlier return of bowel function and shorten the hospital stay, probably via the cephalic-vagal reflex which increase the production of gastrointestinal hormones associated with bowel motility. However, up until now, there has been no strategy or drug that has been consistently effective in accelerating bowel recovery from abdominal surgery.

Coffee is a popular beverage with known influences on the central nervous system and the cardiovascular system. Although coffee can stimulate intestinal function in healthy volunteers, the mechanism by which coffee stimulates intestinal motility is still unknown. The cholinergic anti-inflammatory pathway (CAIP) has been proposed as a key mechanism by which the brain, through the vagus nerve, modulates the immune system in the spleen. Vagal stimulation by nicotine was shown to reduce intestinal inflammation and improve postoperative ileus. It is known that caffeine stimulates vagal activity. An average cup of caffeinated coffee contains 50-150 milligrams of caffeine, depending on the type, concentration and amount of coffee consumed.

The gastrointestinal system can be stimulated by a substantial caloric intake, acidity, osmolality, or volume load. The caloric content of coffee is negligible (approximately 1 kcal/ 100 mL). It has a pH which varies from 5 to 6 (less acidic than other beverages that have no similar effect on the bowel motility). Brewed and filtered coffee is hypotonic (as is water which serves as the control drink in previous studies). Therefore, it seems that the gastrointestinal effect of coffee is most probably not attributed to its physicochemical properties but to the biochemical activity of one or several of the many active compounds in coffee.

In a study that was conducted in 1990, 29% of healthy volunteers claimed that coffee induced a desire to defecate. The effect of caffeinated coffee on recto-sigmoid motor activity was investigated with a manometry. The activity was accelerated four minutes after the intake of either regular or decaffeinated coffee. However, water had no comparable effect on the recto-sigmoid motility. Caffeine, when in the stomach, can act upon gastric myenteric and submucous nerves to induce gastric emptying. The influx of digestive metabolites into the small intestines may stimulate the gastrocolic reflex and be a possible mechanism behind caffeine causing the need to defecate shortly after consumption. The ultimate result of this reflex mediated by caffeine is an increased anal sphincter contraction power and less neural input required to induce contraction (decreased sensory threshold). Rao et al. performed an ambulatory manometry with inserting a catheter through the rectum up to the mid transverse colon. They investigated the effects of 240 mL regular coffee, 240 mL decaffeinated coffee, 240 mL water and a 1000 kcal meal on colonic activity. Regular coffee, decaffeinated coffee and the calorie-rich meal induced more colonic contractions than water. Moreover, regular coffee induced colonic contractions at greater intensity compared to a caloric-rich meal, 60% stronger than water and 23% stronger than decaffeinated coffee. A randomized controlled trial performed in 2012 at the University of Heidelberg among patients after laparoscopic colectomy, studied the effect of coffee on the duration of postoperative ileus. The study showed that the time to first bowel movement was significantly shorter in the group (40 patients) which received 3 caffeinated coffee cups per day compared to group (40 patients) receiving water only. No significant side effects were observed at the active treatment group. Dulskas.A et al. conducted a randomized controlled study in 2015 to evaluate whether consumption of 100 mL coffee is effective in reducing postoperative ileus. The study showed that coffee consumption after colectomy is safe and that decaffeinated coffee was associated with a shorter time to bowel movement and tolerance of solid food but not time to ﬁrst ﬂatus; caffeinated coffee did not impact the duration of postoperative ileus. In all the studies carried out so far, none could explain the mechanism by which coffee stimulates intestinal motility and the determinant agent for this action is still up for discussion: either caffeine or another component of the coffee, such as chlorogenic acids or melanoidins.

Aim The purpose of this study is to evaluate whether the use of caffeine in the post-operative period significantly reduces the duration of postoperative ileus, and therefore, improves recovery and shorten the hospital stay. The study hypothesis is that post-operative use of caffeine will reduce time to recovery of GI function (i.e. reduce post-operative ileus) by at least 15 hours and thus reduce hospital length of stay by at least 15 hours in patients undergoing elective colorectal operations.

Methods This will be a single-centered, prospective, randomized controlled, double blinded trial.

50 patients due to undergo large bowel resection via laparotomy or laparoscopy will be enrolled. Patients will be randomized (1:1) to those who will receive caffeine (study group) and those who will receive placebo (control group). Randomization will occur via an online program (www.randomizer.org) which assigns participants to experimental conditions. Patients in the study group will be given 100 milligrams caffeine citrate orally diluted in 50 milliliters of apple flavored water while patients in the control group will be given 50 milliliters of apple flavored water only. Administration of caffeine or placebo will occur three times per day starting on the morning of postoperative day 1 after surgery until passage of flatus per rectum will occur for the first time or to a maximal period of time of 7 days, whichever comes earlier.

Sample size was calculated as 50 patients (25 pts in each group) which are required in order to have 1-sided α level of 0.05 and a power of 0.80 to detect a difference of 15 hours in the duration of postoperative ileus (standard deviation 21 hours), which is supported by prior studies. Any difference of 15 hours or more between the groups will be statistically significant.

Caffeine or water will be supplied to the surgical floor per participating patient by the pharmacy in coordination with one of the co-investigators who will be un-blinded. At the floor the caffeine or water will be diluted with apple flavored water which will be supplied by the pharmacy, prior to each dose. The investigators (aside from the single un-blinded co-investigator) and primary team of doctors and nurses will be blinded to the patient's assignment.

Postoperative care will be the same for all patients other than the administration of caffeine or placebo. Patients will be instructed to avoid consuming products that contain caffeine (e.g. coffee, tea, chocolate, cola etc.) until the first passage of flatus. No other restrictions on food or beverages consumption will be imposed other than usually are for patients undergoing the same kind of surgery. The patients will be hospitalized under surveillance and monitoring of the primary team during the study period. They will be instructed to keep in mind or to note the endpoints (time to first flatus, time to first bowel movement, time to tolerate solid diet) and to report them to the primary team and study investigators during the routine rounds.

The criteria for hospital discharge include stable vital signs with no febrile morbidity for ≥24 hours, passage of stool, toleration of a regular diet and the absence of other complications.

Safety Endpoints

* Any adverse events deemed possibly, probably or definitely related to treatment with caffeine: arrhythmia, muscle crumps/tremor, restlessness, irritability, headache, dizziness, tachycardia, allergic reactions (rare) or any other severe manifestation that can be attributed to caffeine side effects.
* Any major adverse event resulting from the surgery that might interfere with caffeine or might lead to meaningless endpoint data: organ failure, anastomotic leakage, intraabdominal abscess or invasive re-intervention (Clavien-Dindo classification of surgical complications > 3).

Patients Patients who are scheduled for laparoscopy or open elective colon resection (right or left hemicolectomy, sigmoid resection, anterior resection, segmental colectomy), for an oncologic or inflammatory indication, that are willing to participate in the study will be informed verbally by a member of the study team of the aims, the risks, alternative therapies, their rights and the course of the trial. The investigator will emphasize that study participation is voluntary and the patient can withdraw at any time during the study.

Patients will be included if they fulfill all inclusion criteria and none of the exclusion criteria listed below within the protocol and after written informed consent was obtained. Enrolment period to the study will be 18 months

Statistical analysis Pearson r correlation coefficient will be used to examine the relationship between two Quantitative variables.

T test will be used to compare Quantitative variable between two categories of Qualitative variable.

ANOVA test will be used to compare Quantitative variable between three or more categories of Qualitative variable.

Chi- square test will be used to examine the relationship between two Qualitative variables.

The variables which will be found significantly related to the dependent variable in the monothetic analysis (one-factor-at-a-time method) will be inserted to a multivariate analysis of ANCOVA.

Risks and risk management Most of the population consumes high doses of caffeine (an average coffee consumption of 9-11 kg per person per year) without even noticing. The side effects listed above were previously described after consuming dosages much higher than 3 X 100 mg/day. The safety of caffeine consumption after elective colorectal surgery has been demonstrated through numerous clinical studies as detailed above.

In this study, any patient suffering from a medical condition or requiring treatment with a drug which might interfere with caffeine will be excluded. Therefore, consumption of caffeine in a cumulative dose of 300 mg/day should not cause any side effects.

Despite this, patients will be hospitalized under supervision and monitored by the primary team and study investigators. Documentation of vital signs, physical examination, medical consultants support and assessment of serious adverse events will be conducted. Any unexpected adverse event will be treated efficiently and quickly without extra cost for the patient.

ELIGIBILITY:
Key Inclusion Criteria

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males and females, 18 to 80 years of age inclusive at the time of study screening;
3. Due to undergo large partial / total bowel resection via laparotomy or laparoscopy with primary anastomosis.

Key Exclusion Criteria

1. Scheduled for a colon resection with stoma creation or multi-visceral resection.
2. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures
3. American Society of Anesthesiologists (ASA) Class IV or V
4. History of abdominal carcinomatosis
5. History of radiation enteritis
6. Children <18 or adults > 80 years of age
7. Pregnant women
8. Known allergy to caffeine
9. Consumption of more than 800 milligrams of caffeine (8-10 cups of coffee) daily on a regular basis
10. Complete abstention of caffeine consumption on a regular basis
11. Consumption of drugs which are either substrates or inhibitors of CYP1A2 enzyme (Ciprofloxacin, Fluvoxamine or Clozapine( at the time of the study, due to expected change of caffeine metabolism it these patients
12. Postoperative ventilation, pressor requirement or ICU stay
13. Liver failure or/and liver cirrhosis (MELD>15)
14. Urgent surgery e.g. emergent laparotomy, sepsis, diverting stoma.
15. Opioid treatment for at least a week before surgery.
16. Prior extensive abdominal surgery (not including caesarean section, appendectomy, cholecystectomy or hernia repair).
17. Known impaired mental status or language difficulties.
18. Participation in another interventional trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
First postoperative flatus | Throughout hospital stay for a maximum of 30 days
  The time in hours from end of surgery to first flatus.

SECONDARY OUTCOMES:
First bowel movement | Throughout hospital stay for a maximum of 30 days
  The time in hours from end of surgery to first bowel movement.
Tolerance of solid diet | Throughout hospital stay for a maximum of 30 days
  The time in hours from end of surgery to first solid meal tolerated (the first time the patient is able to eat any food requiring chewing, without vomiting or going back to liquid diet)
Length of postoperative hospital stay. | Throughout hospital stay for a maximum of 30 days
  The postoperative hospital stay is the number of hours from surgery until discharge. The criteria for hospital discharge include stable vital signs with no febrile morbidity for ≥24 hours, passage of stool, toleration of a solid diet and the absence of other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Shussman, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem Region, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H. Postoperative ileus--an update on preventive techniques. Nat Clin Pract Gastroenterol Hepatol. 2008 Oct;5(10):552-8. doi: 10.1038/ncpgasthep1230. Epub 2008 Aug 12. PMID 18695704
- [Background] Basse L, Jakobsen DH, Bardram L, Billesbolle P, Lund C, Mogensen T, Rosenberg J, Kehlet H. Functional recovery after open versus laparoscopic colonic resection: a randomized, blinded study. Ann Surg. 2005 Mar;241(3):416-23. doi: 10.1097/01.sla.0000154149.85506.36. PMID 15729063
- [Background] Jakobsen DH, Sonne E, Andreasen J, Kehlet H. Convalescence after colonic surgery with fast-track vs conventional care. Colorectal Dis. 2006 Oct;8(8):683-7. doi: 10.1111/j.1463-1318.2006.00995.x. PMID 16970579
- [Background] Mattei P, Rombeau JL. Review of the pathophysiology and management of postoperative ileus. World J Surg. 2006 Aug;30(8):1382-91. doi: 10.1007/s00268-005-0613-9. PMID 16850151
- [Background] Wind J, Hofland J, Preckel B, Hollmann MW, Bossuyt PM, Gouma DJ, van Berge Henegouwen MI, Fuhring JW, Dejong CH, van Dam RM, Cuesta MA, Noordhuis A, de Jong D, van Zalingen E, Engel AF, Goei TH, de Stoppelaar IE, van Tets WF, van Wagensveld BA, Swart A, van den Elsen MJ, Gerhards MF, de Wit LT, Siepel MA, van Geloven AA, Juttmann JW, Clevers W, Bemelman WA. Perioperative strategy in colonic surgery; LAparoscopy and/or FAst track multimodal management versus standard care (LAFA trial). BMC Surg. 2006 Nov 29;6:16. doi: 10.1186/1471-2482-6-16. PMID 17134506
- [Background] Asao T, Kuwano H, Nakamura J, Morinaga N, Hirayama I, Ide M. Gum chewing enhances early recovery from postoperative ileus after laparoscopic colectomy. J Am Coll Surg. 2002 Jul;195(1):30-2. doi: 10.1016/s1072-7515(02)01179-1. PMID 12113542
- [Background] George SE, Ramalakshmi K, Mohan Rao LJ. A perception on health benefits of coffee. Crit Rev Food Sci Nutr. 2008 May;48(5):464-86. doi: 10.1080/10408390701522445. PMID 18464035
- [Background] Wu Z, Boersema GS, Jeekel J, Lange JF. Nicotine gum chewing: a novel strategy to shorten duration of postoperative ileus via vagus nerve activation. Med Hypotheses. 2014 Sep;83(3):352-4. doi: 10.1016/j.mehy.2014.06.011. Epub 2014 Jun 17. PMID 24998667
- [Background] Lubbers T, Buurman W, Luyer M. Controlling postoperative ileus by vagal activation. World J Gastroenterol. 2010 Apr 14;16(14):1683-7. doi: 10.3748/wjg.v16.i14.1683. PMID 20379998
- [Background] Hibino G, Moritani T, Kawada T, Fushiki T. Caffeine enhances modulation of parasympathetic nerve activity in humans: quantification using power spectral analysis. J Nutr. 1997 Jul;127(7):1422-7. doi: 10.1093/jn/127.7.1422. PMID 9202101
- [Background] Brown SR, Cann PA, Read NW. Effect of coffee on distal colon function. Gut. 1990 Apr;31(4):450-3. doi: 10.1136/gut.31.4.450. PMID 2338272
- [Background] Conway KJ, Orr R, Stannard SR. Effect of a divided caffeine dose on endurance cycling performance, postexercise urinary caffeine concentration, and plasma paraxanthine. J Appl Physiol (1985). 2003 Apr;94(4):1557-62. doi: 10.1152/japplphysiol.00911.2002. Epub 2002 Dec 13. PMID 12482764
- [Background] Tansy MF, Kendall FM. Experimental and clinical aspects of gastrocolic reflexes. Am J Dig Dis. 1973 Jun;18(6):521-31. doi: 10.1007/BF01076606. No abstract available. PMID 4705102
- [Background] Lohsiriwat S, Kongmuang P, Leelakusolvong S. Effects of caffeine on anorectal manometric findings. Dis Colon Rectum. 2008 Jun;51(6):928-31. doi: 10.1007/s10350-008-9271-y. Epub 2008 Mar 19. PMID 18350336
- [Background] Stacewicz-Sapuntzakis M, Bowen PE, Hussain EA, Damayanti-Wood BI, Farnsworth NR. Chemical composition and potential health effects of prunes: a functional food? Crit Rev Food Sci Nutr. 2001 May;41(4):251-86. doi: 10.1080/20014091091814. PMID 11401245
- [Background] Rao SS, Welcher K, Zimmerman B, Stumbo P. Is coffee a colonic stimulant? Eur J Gastroenterol Hepatol. 1998 Feb;10(2):113-8. doi: 10.1097/00042737-199802000-00003. PMID 9581985
- [Background] Muller S. Author's reply: Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy (Br J Surg 2012; 99: 1530-1538). Br J Surg. 2013 Mar;100(4):573. doi: 10.1002/bjs.9076. No abstract available. PMID 23378207
- [Background] Dulskas A, Klimovskij M, Vitkauskiene M, Samalavicius NE. Effect of Coffee on the Length of Postoperative Ileus After Elective Laparoscopic Left-Sided Colectomy: A Randomized, Prospective Single-Center Study. Dis Colon Rectum. 2015 Nov;58(11):1064-9. doi: 10.1097/DCR.0000000000000449. PMID 26445179
- [Background] Vitaglione P, Fogliano V, Pellegrini N. Coffee, colon function and colorectal cancer. Food Funct. 2012 Sep;3(9):916-22. doi: 10.1039/c2fo30037k. Epub 2012 May 25. PMID 22627289
- [Derived] Parnasa SY, Marom G, Bdolah-Abram T, Gefen R, Luques L, Michael S, Mizrahi I, Abu-Gazala M, Rivkind AI, Mintz Y, Pikarsky AJ, Shussman N. Does caffeine enhance bowel recovery after elective colorectal resection? A prospective double-blinded randomized clinical trial. Tech Coloproctol. 2021 Jul;25(7):831-839. doi: 10.1007/s10151-021-02450-7. Epub 2021 Apr 26. PMID 33900493
- See also: Ref 11. Mayo Clinic staff. Caffeine content for coffee, tea, soda and more. [Accessed March 14, 2017] — http://www.mayoclinic.org/healthy-lifestyle/nutrition-and-healthy-eating/in-depth/caffeine/art-20049372